CLINICAL TRIAL: NCT01810835
Title: Prevention of Hepatitis B Virus (HBV) Mother-to-child Transmission (MTCT): Impact of Serovaccination in Lariboisiere Hospital, Paris, France.
Brief Title: Prevention of Hepatitis B Virus Mother-to-child Transmission by Serovaccination.
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Stephane Mouly, MD PhD, Professor, Medicine A Department, Hopital Lariboisière
Other Study IDs: URT-Liver-001
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis B
Keywords: HBV mother-to-child transmission; women with HBV DNA > 105 I.U./mL; France
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of HBsAg carriage in pregnant women varies in France, according to the native country, with highest rates in those originating from sub-Saharan Africa and Asia (5 to 8 % in Parisian area). The level of HBV-DNA varies according to HBe status and geographical origin, and is strongly predictive of the risk of HBV mother-to-child transmission (MTCT). It has been shown that the rate of vertical transmission (Chinese study by Yuan J et al) was 0 % in newborns to mothers whom HBV-DNA was < 105 copies/mL and up to more than 40 % in newborns to mothers with high viral loads > 108 copies/mL, despite HBIg and vaccine at birth. Thus, data are needed concerning the current practices about the prevention of HBV MTCT in France, and their results.

DETAILED DESCRIPTION:
This monocentre, observational study will include pregnant women whom HBV-DNA is > 105 IU/mL. HBV MTCT rates will be evaluated, according to the level of HBV-DNA in the women during the last three months of pregnancy and at childbirth (between 105 and 108 IU/mL, or > 108 IU/mL), and according to the clinical practices of serovaccination in the participating center. The evaluation will be based on the rate of HBsAg positivity in infants at 9 months, despite a correct immunization at birth. The rate of detectable HBV-DNA will be also evaluated in infants at the same date.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* whom HBs Ag +
* whom HBV-DNA >105 IU/mL

Exclusion Criteria:

* Women who have to be treated for HBV hepatitis, (AST/ALT >2 ULN without any explanation, liver biopsy performed before pregnancy showing hepatitis requiring initiation of treatment)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This monocentre, observational study will include pregnant women whom HBV-DNA is > 105 IU/mL and who are not currently treated for HBV hepatitis.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Rate of HBsAg positivity in infants at 9 months, despite a correct immunization at birth | 9 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O Sellier, M.D., Ph.D., Principal Investigator — Hopital Lariboisiere, Paris, France
Locations (2):
- France (2):
  - Hopital Lariboisiere, Paris
  - Paris